CLINICAL TRIAL: NCT03930446
Title: Alcohol, Behavior, and Brain Imaging
Acronym: (DARC)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB16-0015
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-02

CONDITIONS: Alcohol Drinking; Binge Drinking; Drinking Behavior; Substance-Related Disorders; Ethanol; Physiological Effects of Drugs; Central Nervous System Depressants
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking; Drinking Behavior; Substance-Related Disorders | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ethanol (Experimental): Subjects will receive 4 color-coded beverages in green or blue cups, containing ethanol (0.2 g/kg per dose, total dose 0.8 g/kg).
  Interventions: Drug: Ethanol
- Placebo (Juice) (Placebo Comparator): Subjects will receive 4 color-coded beverages in green or blue cups, containing placebo (Juice).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ethanol — The 0.8 g/kg body weight dose of oral alcohol (190-proof ethanol) will be divided into 4 servings of 0.2 g/kg each. The 0.8 g/kg dose is equivalent to 4 standard drinks, where a standard drink is defined as one 12 oz beer, one 5 oz glass of wine, or one 1.5 oz shot of 80 proof alcohol. Women will receive a reduced dose (0.68 g/kg) to account for sex differences in total body water
  Arms: Ethanol
Other: Placebo — The placebo beverage will consist of the cranberry or orange juice plus 1% alcohol added as a taste mask. All beverages will be sprayed with an alcoholic mist to provide a strong alcoholic scent.
  Arms: Placebo (Juice)

SUMMARY:
To evaluate the relationship of extraversion to both the acute subjective and behavioral effects of alcohol, and the neural reactivity to the anticipation of reward.

ELIGIBILITY:
Inclusion Criteria:

* 21-29 years old
* 7-30 alcoholic drinks per week (as reported on PHQ or TLFB)
* At least one binge episode (4 for females/5 for males) per month
* No 'flushing' reaction to alcohol
* Females must be on birth control or in the beginning of follicular phase (1-14 days after start of menstruation)
* BMI 19-26
* High school education or greater, fluent in English
* No night shift work
* No current or past year Axis I psychiatric disorder including drug/alcohol dependence
* No current psychopharmacological treatment
* No lifetime ADHD or prescription for ADHD medication
* No abnormal EKG, cardiovascular illness, high blood pressure
* No medical condition or pharmacological treatment for which alcohol is contraindicated
* Not pregnant, lactating, or planning to become pregnant
* Smoke <6 cigarettes per day
* No previous participation in studies that have used the Stop Task (except IDAC) o Previous Stop Task studies: GOI, CAP, STEM, JAM, MACI, PAC, CAM

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Weafer, Principal Investigator — University of Chicago

REFERENCES:
- [Derived] Li J, Murray CH, Weafer J, de Wit H. Subjective Effects of Alcohol Predict Alcohol Choice in Social Drinkers. Alcohol Clin Exp Res. 2020 Dec;44(12):2579-2587. doi: 10.1111/acer.14476. Epub 2020 Nov 17. PMID 33201577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ethanol | Placebo (Juice)
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ethanol | Placebo (Juice) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 22 | 22 | 44
  More than one race | 9 | 9 | 18
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Education - High School Education [Count of Participants; unit: Participants] | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Stop Signal Task (SST)
Description: The Stop-Signal Task (SST) is a task requiring inhibition of a prepotent motor response. The SST requires participants to respond to a target stimulus as quickly and accurately as possible by pressing a button, but also to withhold their response when they hear an auditory signal. Thus, this task involves a competition between activating and inhibiting processes. The primary outcome variable is change in the stop signal reaction time (SSRT) for the task administered seconds to minutes before and seconds to minutes after stimulation. The theoretical minimum is zero seconds and there is no theoretical maximum. Higher SSRT scores reflect greater impulsivity.
Time Frame: Within an hour post-stimulation condition
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Ethanol | Placebo (Juice)
Number analyzed (Participants) | 40 | 40
milliseconds | 255 (463) | 215 (278)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 weeks
Arm/Group | Ethanol | Placebo (Juice)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT03930446/Prot_SAP_000.pdf